CLINICAL TRIAL: NCT03174301
Title: Prematurity-Related Ventilatory Control: Role in Respiratory Outcomes
Acronym: Pre-Vent
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: Case Western Reserve University (Other); Northwestern University (Other); University of Alabama at Birmingham (Other); University of Miami (Other); Washington University School of Medicine (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Brown University (Other)
Responsible Party: Principal Investigator, Joseph R Moorman, Professor of Medicine, University of Virginia
Other Study IDs: 19606; U01HL133708 (NIH)
Record Dates: First submitted 2017-05-19; First posted 2017-06-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Infant, Premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this common multicenter protocol is to test the hypothesis that algorithmic tools using clinical Neonatal Intensive Care Unit (NICU) cardiorespiratory monitoring data can detect ventilatory control instability and predict chronic and acute respiratory consequences of ventilatory control instability and autonomic dysregulation.

ELIGIBILITY:
Inclusion Criteria:

* Neonatal Intensive Care Unit patient on cardiorespiratory monitor which has been configured to collect data to store for this study
* < 29 wks Gestational Age
* < 1 wk Chronological

Exclusion Criteria:

* Unlikely to survive or decision not to pursue full care
* Major congenital or chromosomal anomaly

Max Age: 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All races and ethnicities will be recruited and distribution is expected to be similar to the populations represented in the NICU at each site.
  Age of all infants will be less than 29 weeks Gestational Age and less than 1 week Chronological Age, at the time of enrollment.
  The study population will be drawn from inpatients in NICUs at participating hospital sites with cardiorespiratory monitoring.
  The subjects will be in variable states of health since they are premature and in the intensive care unit.
  There will be no pre-screening of infants. Data will be collected on all infants placed in a bed for which monitoring and data collection capabilities are set up. Therefore all such infants will technically be enrolled in the study, regardless of meeting the inclusion/exclusion criteria.
  Each enrolled infant will be screened for inclusion/exclusion criteria to determine whether the site will collect further data from the medical record.
Sampling Method: Non-Probability Sample
Enrollment: 739 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Clinical Outcome | 40 weeks post-menstrual age.
  "Favorable": Either (1) an inpatient at 40 weeks post-menstrual age and not on oxygen, nor on other flow/pressure respiratory support, nor on inhaled/oral/IV respiratory medications, OR (2) discharged prior to 40 weeks post-menstrual age not on respiratory meds, oxygen, or other respiratory support.
  "Unfavorable": Either (1) Deceased at 40 weeks , (2) inpatient on meds/O2/support at 40 weeks post-menstrual age, or (3) previously discharged prior to 40 weeks on meds/O2/support
Physiological Outcome | 36 weeks and 1 day to 37 weeks and 0 days, post-menstrual age
  Reported Value will be the percentile value of scores, as plotted on a standard curve of scores for peers. The score is calculated by aggregating the following measurements:
  1. Periodic Breathing Percentage (%)
  2. Number of Apnea events (#)
  3. Number of Bradycardia events (#)
  4. Number of Desaturation events (#)
  5. Number of combined events (example Apnea with Bradycardia and Desaturation (#)

SECONDARY OUTCOMES:
time on respiratory support and medications | before 52 weeks post-menstrual age
chronic lung disease | before 52 weeks post-menstrual age
pulmonary hypertension | before 52 weeks post-menstrual age
sepsis | before 52 weeks post-menstrual age
necrotizing enterocolitis | before 52 weeks post-menstrual age

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and linked DNA samples will be stored at NHLBI Biorepository BIO-LINCC. Data will include continuous cardio-respiratory monitoring, demographics, clinical events, co-morbidities, respiratory status, and other clinical data.

REFERENCES:
- [Derived] Travers CP, Chahine R, Nakhmani A, Aban I, Carlo WA, Ambalavanan N. Control of breathing in preterm infants on incubator oxygen or nasal cannula oxygen. Pediatr Res. 2025 Feb;97(3):1166-1170. doi: 10.1038/s41390-024-03460-5. Epub 2024 Aug 15. PMID 39147903
- [Derived] Kausch SL, Lake DE, Di Fiore JM, Weese-Mayer DE, Claure N, Ambalavanan N, Vesoulis ZA, Fairchild KD, Dennery PA, Hibbs AM, Martin RJ, Indic P, Travers CP, Bancalari E, Hamvas A, Kemp JS, Carroll JL, Moorman JR, Sullivan BA; Prematurity-Related Ventilatory Control (Pre-Vent) Investigators. Apnea, Intermittent Hypoxemia, and Bradycardia Events Predict Late-Onset Sepsis in Infants Born Extremely Preterm. J Pediatr. 2024 Aug;271:114042. doi: 10.1016/j.jpeds.2024.114042. Epub 2024 Apr 2. PMID 38570031
- [Derived] Kausch SL, Lake DE, Di Fiore JM, Weese-Mayer DE, Claure N, Ambalavanan N, Vesoulis ZA, Fairchild KD, Dennery PA, Hibbs AM, Martin RJ, Indic P, Travers CP, Bancalari E, Hamvas A, Kemp JS, Carroll JL, Moorman JR, Sullivan BA; Prematurity-Related Ventilatory Control (Pre-Vent) Investigators. Apnea, Intermittent Hypoxemia, and Bradycardia Events Predict Late-Onset Sepsis in Extremely Preterm Infants. medRxiv [Preprint]. 2024 Jan 27:2024.01.26.24301820. doi: 10.1101/2024.01.26.24301820. PMID 38343825